CLINICAL TRIAL: NCT06544343
Title: Integration of Remote Monitoring in the Management of Chronic Immunosuppressive Therapy in Patients With Rheumatologic Diseases: Comparison With Standard Management
Brief Title: Integration of Remote Monitoring in the Management of Chronic Immunosuppressive Therapy
Acronym: TEMPLATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Elena Bartoloni Bocci, Associate Professor, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4663/24
Record Dates: First submitted 2024-07-19; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Systemic Lupus Erythematosus; Systemic Sclerosis; Spondyloarthritis, Axial; Ankylosing Spondylitis
Keywords: Immunosuppression; Quality of Life
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Axial Spondyloarthritis; Spondylitis, Ankylosing | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Monitoring (Experimental)
  Interventions: Other: Remote Monitoring; Other: On site monitoring
- On site only (Placebo Comparator)
  Interventions: Other: On site monitoring

INTERVENTIONS:
Other: Remote Monitoring — Follow-up at outpatient clinic at 3 and 6 months from drug prescription Two remote consultations at 15 and 45 days from drug prescription
  Arms: Remote Monitoring
Other: On site monitoring — Follow-up at outpatient clinic at 3 and 6 months from drug prescription.

SUMMARY:
Systemic autoimmune and chronic inflammatory diseases are a group of chronic illnesses whose treatment is usually very prolonged, often lifelong, and is essential to keep the disease under control, thus reducing the risk of complications and allowing the best possible quality of life for patients.

The drugs used for treating these diseases are mostly immunosuppressants, which reduce the activity of the immune system, whose alteration is responsible for the disease. Although all available drugs are effective for treating these diseases, for reasons largely unknown, each drug is effective only in a percentage of patients. As a result, it is often necessary to try several different treatments before identifying an effective one for the individual patient.

The therapeutic effects are often slow, and it is therefore necessary to take a treatment for weeks or months before its effectiveness can be determined. The initial period is also when side effects most often appear. The aim of this study is to evaluate whether the addition of remote monitoring visits and other patient support services to traditional periodic medical visits in the first months after the introduction of a new treatment leads to an improvement in adherence, response, and quality of life for the patient.

ELIGIBILITY:
Inclusion Criteria:

Any patient with one of the following conditions

* Rheumatoid Arthritis
* Psoriatic Arthritis
* Spondyloarthritis
* Ankylosing Spondylitis
* Systemic Sclerosis
* Systemic Lupus Erythematosus
* Sjogren's Disease who are prescribed a new immunosuppressive medication for the treatment of their disease among the following:
* Methotrexate
* Sulfasalazine
* Leflunomide
* Mycophenolate Mofetil
* Azathioprine
* Cyclosporine A
* Tacrolimus
* TNF inhibitors (etanercept, adalimumab, golimumab, certolizumab pegol)
* IL6 inhibitors (tocilizumab)
* IL-17 inhibitors (secukinumab, ixekizumab)
* IL-23 inhibitors (ustekinumab, guselkumab, risankizumab)
* JAK-inhibitors (tofacitinib, baricitinib, upadacitinib, filgotinib)
* Belimumab
* Anifrolumab

Exclusion Criteria:

* Treatment with a medication not approved for the condition
* Inability to use a device for remote call, not even with the help of a caregiver

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Treatment persistence | 6 months
  Percentage of patients taking the same medication prescribed at baseline

SECONDARY OUTCOMES:
Treatment Persistence | 3 months
  Percentage of patients taking the same medication prescribed at baseline
Disease activity score on 28 joints with C-Reactive Protein (DAS28-CRP) | 3 months
  Only applies to rheumatoid arthritis patients
Disease activity score on 28 joints with C-Reactive Protein (DAS28-CRP) | 6 months
  Only applies to rheumatoid arthritis patients
Psoriatic Arthritis Disease Activity Score (PASDAS) | 3 months
  Only applies to psoriatic arthritis patients
Psoriatic Arthritis Disease Activity Score (PASDAS) | 6 months
  Only applies to psoriatic arthritis patients
Body Surface Area (BSA) | 3 months
  Percentage of skin surface with psoriatic lesions. Only applies to psoriatic arthritis patients
Body Surface Area (BSA) | 6 months
  Percentage of skin surface with psoriatic lesions. Only applies to psoriatic arthritis patients
Minimal Disease Activity (MDA) | 3 months
  Binary outcome. Only applies to psoriatic arthritis patients
Minimal Disease Activity (MDA) | 6 months
  Binary outcome. Only applies to psoriatic arthritis patients
Modified Rodnan's skin score | 3 months
  Only applies to systemic sclerosis patients
Modified Rodnan's skin score | 6 months
  Only applies to systemic sclerosis patients
Medical Research Council (MRC) dyspnoea scale | 3 months
  Only applies to systemic sclerosis patients with interstitial lung disease
Medical Research Council (MRC) dyspnoea scale | 6 months
  Only applies to systemic sclerosis patients with interstitial lung disease
EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) | 3 months
  Only applies to Sjogren's disease patients
EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) | 6 months
  Only applies to Sjogren's disease patients
EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) | 3 months
  Only applies to Sjogren's disease patients
EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) | 6 months
  Only applies to Sjogren's disease patients
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K | 3 months
  Only applies to systemic lupus erythematosus patients
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)-2K | 6 months
  Only applies to systemic lupus erythematosus patients
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 3 months
  Only applies to ankylosing spondylitis and axial spondyloarthritis patients
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 6 months
  Only applies to ankylosing spondylitis and axial spondyloarthritis patients
Health Assessment Questionnaire Disability Index (HAQ-DI) | 3 months
  Range 0 (best condition) - 3 (worst condition)
Health Assessment Questionnaire Disability Index (HAQ-DI) | 6 months
  Range 0 (best condition) - 3 (worst condition)
Anxiety and Depression | 3 months
  Hospital Anxiety and Depression Scale - Anxiety and Depression range 0 - 21 each (higher values mean higher degrees of depression or anxiety)
Anxiety and Depression | 6 months
  Hospital Anxiety and Depression Scale - Anxiety and Depression range 0 - 21 each (higher values mean higher degrees of depression or anxiety)
EQ-5D-5L score | 3 months
  The score measures quality of life and includes 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which is scored from 1 (perfect health) to 5 (complete inability).
EQ-5D-5L score | 6 months
  The score measures quality of life and includes 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which is scored from 1 (perfect health) to 5 (complete inability).
Number of phone calls to Rheumatology Outpatient Clinic | 6 months
Number of additional, unscheduled rheumatology consultations | 6 months
Number of consultations to GP due to prescribed treatment-related issues | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Unit - Perugia Univeristy Hospital, Perugia, PG, Italy

IPD SHARING:
Plan to Share IPD: No